CLINICAL TRIAL: NCT03530332
Title: Prediction and Prevention of Preterm Birth: A Prospective, Randomized Intervention Trial
Brief Title: Prediction and Prevention of Preterm Birth (PREVENT-PTB Study)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inadequate resources.
Sponsor: Ware Branch (Other)
Collaborators: Sera Prognostics, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Ware Branch, Medical Dir Sr - Women/Newborn, Intermountain MFM Specialist, Intermountain Health Care, Inc.
Organization: Intermountain Health Care, Inc. (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PREVENT-PTB Protocol 1.02
Record Dates: First submitted 2018-05-08; First posted 2018-05-21 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Preterm Birth
Keywords: Preterm Birth; Prematurity Prevention Clinic; Maternal-Fetal Medicine
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Experimental)
  Interventions: Diagnostic Test: PreTRM test
- Control (No Intervention)

INTERVENTIONS:
Diagnostic Test: PreTRM test — Blood test to determine risk of preterm birth
  Arms: Treatment

SUMMARY:
This research study is being done to find out whether a screening blood test can help identify women with an increased risk of preterm birth.

DETAILED DESCRIPTION:
Preterm birth (PTB) remains the leading cause of neonatal mortality and long-term disability throughout the world. Recently treatments early in pregnancy such as progesterone, cervical support and maternal support have been demonstrated to delay delivery amongst at risk women. Nonetheless, the majority of women who are at risk are not identified using current screening methods.

Women who are 18 years or older, with a singleton pregnancy between 19 5/7 weeks and 20 6/7 weeks gestational age (GA) confirmed by ultrasound prior to enrollment and no history of prior preterm birth (delivery between 16 0/7 weeks and 37 6/7 weeks) will be invited to participate. Women who enroll will be randomized to screening and intervention for those at high risk of PTB or no screening and standard care. All participants will undergo sample collection, but the samples from the group randomized to "no screening' will not be analyzed until the end of the study (post-delivery of all neonates).

Women randomized to the intervention group will be screened using the PreTRM® test (Sera Prognostics, Inc.) at a large tertiary care center. Predicated upon the degree of risk, women will be treated according to a pre-specified algorithm. The outcomes of these women will be compared to a control group of women who do not receive screening at the same tertiary care center.

ELIGIBILITY:
Inclusion Criteria

1. Subject is greater than or equal to 18 years of age AND
2. Uncomplicated singleton intrauterine pregnancy less than 21 weeks estimated gestation AND
3. No medical contraindications to continuing pregnancy AND
4. No previous classical cesarean section AND
5. No known uterine anomaly AND
6. No history of cervical conization AND
7. No plan for cesarean section prior to 37 0/7 weeks gestation AND
8. No plan for induction of labor prior to 37 0/7 weeks gestation AND
9. Subject has no history of spontaneous preterm delivery AND
10. No prior PPROM less than 34 weeks AND
11. Subject has no signs and/or symptoms of preterm labor AND
12. Subject has intact membranes AND
13. Subject has not received a blood transfusion during the current pregnancy.

Exclusion Criteria

1. Subjects who have taken or plan to take progesterone beyond 13 6/7 weeks gestation prior to study enrollment OR
2. Any other medical conditions that put subject at increased risk of preterm birth in the judgment of the site investigator OR
3. The subject has a planned cerclage placement for the current pregnancy OR
4. Previously identified short cervix (less than 2.5 cm by transvaginal ultrasound) prior to enrollment OR
5. Known major structural fetal anomalies that may shorten pregnancy (e.g., anencephaly, holoprosencephaly, schizencephaly, gastroschisis, omphalocele, congenital diaphragmatic hernia) OR
6. Known fetal genetic anomalies that are incompatible with life (e.g., trisomy 13 or trisomy 18) OR
7. The subject has known elevated bilirubin levels (hyperbilirubinemia) OR
8. The subject has taken or plans to take any of the following medications after the first day of the last menstrual period: Enoxaparin, heparin, heparin sodium, low molecular weight heparin, low dose aspirin OR
9. A history of allergic reaction to aspirin or 17-OHPC injections OR
10. Subject does not plan to deliver at an Intermountain Healthcare hospital.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1208 (Actual)
Dates: Start 2018-05-14 (Actual); Primary Completion 2019-02-17 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Incidence of spontaneous preterm birth | Before 37 weeks of pregnancy

SECONDARY OUTCOMES:
Gestational age at delivery | At delivery
Neonatal Intensive Care Unit (NICU) length of stay only among neonates who were admitted to the NICU | Up to 1 year post delivery
Length of stay among all neonates (including NICU and nursery) | Up to 1 year post delivery
Neonatal costs | Up to 1 year post delivery

CONTACTS AND LOCATIONS:
Overall Officials: Ware Branch, M.D., Principal Investigator — Intermountain Health Care, Inc.
Locations (4):
- United States (4):
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital, Ogden, Utah
  - Utah Valley Hospital, Provo, Utah
  - LDS Hospital, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Branch DW, VanBuren JM, Porter TF, Holmgren C, Holubkov R, Page K, Burchard J, Lam GK, Esplin MS. Prediction and Prevention of Preterm Birth: A Prospective, Randomized Intervention Trial. Am J Perinatol. 2023 Jul;40(10):1071-1080. doi: 10.1055/s-0041-1732339. Epub 2021 Aug 16. PMID 34399434